CLINICAL TRIAL: NCT01747642
Title: Study to Evaluate Safety and Therapeutic Efficacy of a Combination Therapy of 'Oncoxin', a Nutritional Supplement and Surafenib, a Multikinase Inhibitor in Patients With Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Oncoxin Plus Surafineb in Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Organization, Dhaka, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP2
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Quality of Life
Keywords: Hepatocellular carcinoma; Oncoxin; Surafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oncoxin (Active Comparator): Syp Oncoxin 25 ml bd and Cap. Oncoxin bd orally for 180 days
  Interventions: Dietary Supplement: Oncoxin
- Oncoxin & Suranix (Active Comparator): Tab Suranix 200 mg 2 tab bd and Syp Oncoxin 25 ml bd and Cap. Oncoxin bd orally for 180 days
  Interventions: Dietary Supplement: Oncoxin; Drug: Suranix
- Supportive treatment (No Intervention): Only supportive treatment. No chemotherapy, radoiotherapy, ablation or surgical intervention will be carried out.

INTERVENTIONS:
Dietary Supplement: Oncoxin — Syp Oncoxin 25 ml bd and Cap. Oncoxin bd for 180 days
  Arms: Oncoxin; Oncoxin & Suranix
Drug: Suranix — Tab Suranix 200 mg 2 tab bd and Syp Oncoxin 25 ml bd and Cap. Oncoxin bd for 180 days
  Other Names: Nexavar; Suranib
  Arms: Oncoxin & Suranix

SUMMARY:
Oncoxin in combination with Surafenib is safe and results in improved survival in patients with hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
To assess therapeutic efficacy and safety of Oncoxin plus Surafenib in hepatocellular carcinoma

To see if there is reduction in serum alpha fetoprotein level in hepatocellular carcinoma patients after administration of Oncoxin plus Surafenib

To see if there is reduction tumor size and or number in hepatocellular carcinoma patients after administration of Oncoxin plus Surafenib

To see if there is improvement of quality of life in hepatocellular carcinoma patients after administration of Oncoxin plus Surafenib

To see if there is improved survival in hepatocellular carcinoma patients after administration of Oncoxin plus Surafenib

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC irrespective of etiology, age, gender and status of underlying liver disease.
* Patients with HCC who are not suitable candidates for established modalities of treatment i.e. surgery and/or chemotherapy.
* Patients with HCC who have evidence of tumor metastasis
* Patients with HCC who are voluntarily unwilling to take established modalities of treatment i.e. surgery and/or chemotherapy.
* Patients with HCC in whom all possible treatment options have been exhausted.

Exclusion Criteria:

* Patients with HCC who are suitable candidates for established modalities of treatment i.e. surgery and/or chemotherapy.
* Patients with HCC who have no evidence of tumor metastasis
* Patients with HCC who are willing to take established modalities of treatment i.e. surgery and/or chemotherapy.
* Patients with HCC who are voluntarily unwilling to be included in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have prolonged survival | 24 weeks
  To study the number of participants who have prolonged survival in months after receiving Oncoxin plus Surafenib for 24 weeks

SECONDARY OUTCOMES:
Reduction in serum alpha-fetoprotein level and decrease in tumor size | 24 weeks
  To see whether Oncoxin plus Surafenib results in reduction in serum alpha-fetoprotein level in ng/ml and decrease in tumor size in mm in hepatocellular carcinoma patients off treatment for 24 weeks, after receiving Oncoxin plus Surafenib for 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mamun A Mahtab, MD, FACG, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Farabi General Hospital, Dhaka, Bangladesh